CLINICAL TRIAL: NCT02814357
Title: To Evaluate the Effect of 4 Different Flour Compositions of Selected Fibres and Flours, on Post-prandial Plasma Glucose (PPG) and Serum Insulin Levels in Normal Indian Healthy Subjects
Brief Title: To Test the Effect of Selected Fibres and Flours in Flat Bread on Post-Prandial Blood Glucose and Insulin Responses in Healthy Indian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FDS-NAA-0224
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: Blood glucose, serum insulin
MeSH Terms: interventions — Flour; guar gum

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (market standard) (Placebo Comparator): 100 g wheat flour (atta)
  Interventions: Other: Control (market standard)
- High fibre 1 (Active Comparator): 81% wheat flour (atta) + 15% chickpea + 4% guar gum
  Interventions: Other: wheat flour; Other: chickpea flour; Other: guar gum
- High fibre 2 (Active Comparator): 80% wheat flour (atta) + 15% chickpea + 2% guar gum + 3% barley
  Interventions: Other: wheat flour; Other: chickpea flour; Other: guar gum; Other: barley
- High fibre 3 (Active Comparator): 77% wheat flour (atta) + 15% chickpea + 3% guar gum + 5% barley
  Interventions: Other: wheat flour; Other: chickpea flour; Other: guar gum; Other: barley

INTERVENTIONS:
Other: Control (market standard)
  Arms: Control (market standard)
Other: wheat flour
  Arms: High fibre 1; High fibre 2; High fibre 3
Other: chickpea flour
  Arms: High fibre 1; High fibre 2; High fibre 3
Other: guar gum
  Arms: High fibre 1; High fibre 2; High fibre 3
Other: barley
  Arms: High fibre 2; High fibre 3

SUMMARY:
Double-blind, randomized, controlled, cross-over design with 3 test products and one control product.

To evaluate the effect of 4 different flour compositions (guar gum 2% and 4%, chickpea flour 15% and barley flour 2% and 5%) of selected fibres and flours, on post-prandial plasma (PPG) and serum insulin levels in healthy Indian subjects, after the consumption of flat bread made from 100 gram of flour compositions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between > 20 and < 50 years of age
* BMI of >18 and < 23 kg/m2
* Fasting blood glucose value of volunteer is > 3.4 and <6.1 mmol/litre (i.e. 62- 110 mg/dl) at screening

Exclusion Criteria:

* Chronic smokers, tobacco chewers and drinkers.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Positive incremental area under blood glucose curve | 0-120 minutes

SECONDARY OUTCOMES:
Total area under the serum insulin curve | 0-120 minutes

OTHER OUTCOMES:
Cmax glucose | 0-120 minutes
Tmax glucose | 0-120 minutes
Slope to Cmax | 0-120 minutes
Glucose concentration | 180 minutes
Insulin concentration | 180 minutes
Total area under the glucose curve | 0-180 minutes
Total area under the curve of appetite and mood | 0-120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Patel, Dr., Principal Investigator — Lambda Therapeutic Research Ltd.
Locations (1):
- Lambda Therapeutics Research Ltd (LTRL), Ahmedabad, Near Gujrat High Court, SG Highway, Gota, India